CLINICAL TRIAL: NCT02373982
Title: External Validation of the Left Atrial Sphericity as Predictor of Recurrence After Atrial Fibrillation Ablation: A Multicenter Observational Study.
Brief Title: Left Atrial Geometry and Outcomes After Atrial Fibrillation Ablation
Acronym: LAGO-FA
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital del Mar (Other); Hospital Virgen de la Salud (Other); Hospital San Carlos, Madrid (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); Complejo Hospitalario Universitario de Vigo (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, MD, PhD, FESC, Hospital Clinic of Barcelona
Other Study IDs: LAGO-FA
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Multicenter Observational 1-year retrospective cohort study evaluating the predictive value of the Left Atrial Sphericity on the recurrence rate of atrial fibrillation after pulmonary vein ablation procedure.

Inclusion of consecutive patients undergoing AF ablation during 2013 in whom a 3D-imaging of the left atrium (Cardiac CT or MRA) was acquired prior to the procedure and when procedural/follow-up data was prospectively collected.

DETAILED DESCRIPTION:
Validation of the predictive value of the Left Atrial Sphericity for AF recurrence of atrial fibrillation after a pulmonary vein ablation procedure in an external, multicenter cohort.

In total, 9 centers will include consecutive patients who underwent AF ablation from january to december 2013 in whom a 3D-imaging of the left atrium (Cardiac CT or MRA) was acquired prior to the procedure and when procedural/follow-up data was prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* First AF ablation procedure
* Prior 3D-imaging of the left atrium (CT or MRA)
* Prospective collection procedural and outcome data
* Obtention of Informed Consent

Exclusion Criteria:

* Previous left atrial ablation or surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-center cohort of consecutive patients undergoing first ablation of symptomatic drug-refractory AF during 2013 in whom 3D-imaging of the left atrium was performed (Cardiac CT or MRA).
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Recurrence (>30 seconds) | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Bisbal, MD, Principal Investigator — Germans Trias i Pujol Hospital; Lluís Mont, MD PhD, Principal Investigator — Hospital Clinic
Locations (9):
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clinico de Valencia, Valencia
  - Complexo Hospitalario de Vigo, Vigo

REFERENCES:
- [Background] Bisbal F, Guiu E, Calvo N, Marin D, Berruezo A, Arbelo E, Ortiz-Perez J, de Caralt TM, Tolosana JM, Borras R, Sitges M, Brugada J, Mont L. Left atrial sphericity: a new method to assess atrial remodeling. Impact on the outcome of atrial fibrillation ablation. J Cardiovasc Electrophysiol. 2013 Jul;24(7):752-9. doi: 10.1111/jce.12116. Epub 2013 Mar 14. PMID 23489827
- [Background] Bisbal F, Guiu E, Cabanas P, Calvo N, Berruezo A, Tolosana JM, Arbelo E, Vidal B, de Caralt TM, Sitges M, Brugada J, Mont L. Reversal of spherical remodelling of the left atrium after pulmonary vein isolation: incidence and predictors. Europace. 2014 Jun;16(6):840-7. doi: 10.1093/europace/eut385. Epub 2014 Jan 2. PMID 24390389
- [Background] Steinberg BA, Piccini JP. Left atrial remodeling: shape before size? J Cardiovasc Electrophysiol. 2013 Jul;24(7):760-1. doi: 10.1111/jce.12132. Epub 2013 Apr 9. No abstract available. PMID 23574013
- [Derived] Bisbal F, Alarcon F, Ferrero-de-Loma-Osorio A, Gonzalez-Ferrer JJ, Alonso C, Pachon M, Tizon H, Cabanas-Grandio P, Sanchez M, Benito E, Teis A, Ruiz-Granell R, Perez-Villacastin J, Vinolas X, Arias MA, Valles E, Garcia-Campo E, Fernandez-Lozano I, Villuendas R, Mont L. Left atrial geometry and outcome of atrial fibrillation ablation: results from the multicentre LAGO-AF study. Eur Heart J Cardiovasc Imaging. 2018 Sep 1;19(9):1002-1009. doi: 10.1093/ehjci/jey060. PMID 29659784